CLINICAL TRIAL: NCT06274814
Title: Ultrasound Guided Rhomboid Intercostal Block Combined With Sub-Serratus Plane Block vs Type 2 Pectoral Nerve Block in Analgesia for Breast Cancer Surgery
Brief Title: U/S Guided Rhomboid Intercostal Block Combined With Sub-Serratus Plane Block vs Type 2 Pectoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Soliman, lecturer of anesthesia, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AP23.501.038
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Breast Neoplasm Female; Analgesics
Keywords: Analgesics; Opioids; Breast Neoplasms; Postoperative Pain; Mastectomy; Nerve block; Breast Cancer Surgery
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type 2 Pectoral Nerve Block (Active Comparator): 23 patients Type 2 Pectoral Nerve Block pecs2 Group A
  Interventions: Procedure: U/S guided Type 2 Pectoral Nerve Block
- RISS Rhomboid intercostal block combined with the sub-serratus plane block (Active Comparator): 23 patients the RIB combined with the sub-serratus plane block (RISS) Group B
  Interventions: Procedure: U/S guided RIB combined with the sub-serratus plane block (RISS)
- No block intervention (No Intervention): routine IV analgesia 23 patients no block intervention was performed. The anesthetic dose was adjusted to maintain blood pressure within 20% of the baseline value. An additional dose of intravenous fentanyl (0.1 µg kg-1 min-1) was injected as needed.
  Group C

INTERVENTIONS:
Procedure: U/S guided Type 2 Pectoral Nerve Block — 20 mL separates the pectoralis major and minor muscles, while 10 mL separates the serratus and pectoralis major muscles
  Arms: Type 2 Pectoral Nerve Block
Procedure: U/S guided RIB combined with the sub-serratus plane block (RISS) — he ipsilateral arm was abducted. RISS was performed. Using a 6-13 MHz linear ultrasound probe was placed medial to the medial border of the scapula in the oblique sagittal plane.. A 100-mm 21-gauge needle was inserted at the level of T5-6 in the ultrasound view. A single dose of 20-mL 0.25% bupivacaine was injected in the interfascial plane between the rhomboid major and intercostal muscles. The spread of the local anesthetic solution under the rhomboid muscle was visualized by ultrasonography. Thereafter, the ultrasound probe was moved caudally and laterally to identify the tissue plane between the serratus anterior and external intercostal muscles for the sub-serratus block at the T8-9 level. The needle was advanced from its previous position, and an additional 20 mL of 0.25% bupivacaine was injected.
  Arms: RISS Rhomboid intercostal block combined with the sub-serratus plane block

SUMMARY:
The aim of this study is to compare between U/S Guided Rhomboid Intercostal Block Combined with Sub-Serratus Plane Block vs type 2 Pectoral Nerve Block in Analgesia for Breast Cancer Surgery by measuring intraoperative hemodynamics, postoperative pain scores and morphine consumption in the first 24 h postoperative.

DETAILED DESCRIPTION:
Patients will be randomly allocated into three groups based on a computerized randomization table with specific ID for each patient (23 per group). Each patient will be prepared in Preoperative Holding Area with sedation with midazolam 0.05mg/kg patients allotted to the RIB group were positioned in the lateral decubitus position with the breast on the operating side lying superiorly. The ipsilateral arm was abducted from the chest to move the scapula laterally. The RISS was performed after application of antiseptic solution. A high-frequency using a 6-13 MHz linear ultrasound probe set to B mode (SonoSite M-turbo ultrasound machine) was placed medial to the medial border of the scapula in the oblique sagittal plane. The landmarks, i.e., the trapezius muscle, rhomboid muscle, intercostal muscles, pleura, and lung, were identified in the ultrasound. Under aseptic conditions, a 100-mm 21-gauge needle was inserted at the level of T5-6 in the ultrasound view. A single dose of 20-mL 0.25% bupivacaine was injected in the interfascial plane between the rhomboid major and intercostal muscles. The spread of the local anesthetic solution under the rhomboid muscle was visualized by ultrasonography. Thereafter, the ultrasound probe was moved caudally and laterally to identify the tissue plane between the serratus anterior and external intercostal muscles for the sub-serratus block at the T8-9 level. The needle was advanced from its previous position, and an additional 20 mL of 0.25% bupivacaine was injected. All block procedures were performed by the same anesthesiologist who had administered the RIB and RISS blocks in more than 30 cases before this study. In control group (Group C), no block intervention was performed.

After disinfection, using 30 mL of levobupivacaine 0.25% (10 mL between pectoralis minor muscle and pectoralis major muscle, and 20 mL between the pectoralis major muscle and serratus muscle). With the patient in supine position. (Group B) After shifting to the operative area, all patients underwent conventional monitoring procedures including electrocardiography, noninvasive monitoring of blood pressure, and peripheral oxygen saturation measurements. Intravenous access was gained using a 22-gauge intravenous needle, and isotonic saline was infused at a rate of 15 mL kg-1 h-1. Anesthetic management was in accordance with a standard protocol. Anesthesia was induced with pre-oxygenation for 3 min followed by intravenous injection of midazolam (0.05 mg/kg), fentanyl (0.1 µg/kg), propofol (1-2 mg/kg), and atracurium (0.5 mg/kg). An endotracheal tube was used for positive-pressure ventilation to maintain the end-tidal carbon dioxide level of 35-40 mmHg.

Anesthesia was maintained using 2% sevoflurane with 50% oxygen, fentanyl (0.1 µg kg-1 min-1), and propofol (100 µg kg-1 min-1). Additionally, atracurium (0. 1 mg/kg) was administered according to the surgical protocol. Surgery (Unilateral conservative mastectomy) was started. The anesthetic dose was adjusted to maintain blood pressure within 20% of the baseline value. An additional dose of intravenous fentanyl (0.1 µg kg-1 min-1) was injected as needed. If the blood pressure decreased by > 20% from the baseline value, 250 mL of 0.9% (physiologic) saline and ephedrine (0.1 mg/kg) were administered. If the heart rate decreased to less than 50 bpm, atropine (0.5 mg/kg) was administered. At the end of the surgery, the effect of atracurium was reversed using neostigmine and atropine as needed. After the surgery, the endotracheal tube was removed when the patient fulfills criteria of extubation. Then the patient will be transferred to the PACU.

Data will be collected:

A. Intraoperative assessment: (readings will be taken just after induction and every 15 min throughout surgery)

1. Heart rate intraoperative.
2. Mean arterial blood pressure intraoperative.
3. Analgesic consumption: recorded during intraoperative period to maintain maximum 20% change of basal vital signs after exclusion of other causes. (Intraoperative fentanyl consumption)

B. Postoperative:

1. Recovery time: the time taken to be fully awake and responding to commands.
2. Pain score: VAS score at 0, 3, 6, 9,24h post-operative.
3. Hemodynamic: pulse, B.P (systolic, diastolic, and mean blood pressure) at 0,3,6,9,24h postoperative.
4. Side effects (nausea, vomiting, hematoma, hypotension, bradycardia).
5. Rescue analgesia plane will be given for VAS≥4 using non-steroidal anti-inflammatory analgesic (ketorolac 30 mg) and VAS≥6 using opioid (3mg morphine). Time of the first rescue analgesia together with frequency and total dose of the given drug through the 24 hours will be recorded.
6. Hospital discharge.

Primary outcome:

1. Total morphine consumption in first 24 hours post operative.
2. VAS score postoperative.

Secondary outcome:

1. Heart rate intraoperative.
2. Mean arterial blood pressure intraoperative.
3. Timing of first rescue analgesia.
4. Intraoperative fentanyl consumption.
5. Side effects (nausea, vomiting, hematoma, hypotension, bradycardia).
6. Body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients.
2. Scheduled for unilateral conservative mastectomy.
3. Age 18-65 years.
4. American Society of Anesthesiologists (ASA) physical status I- II.

Exclusion Criteria:

1. Patient refusal.
2. Coagulation disorders.
3. Body mass index > 40 kg/m2.
4. Uncooperative or psychiatric patients.
5. Infection at the injection site.
6. Patients with a history of allergy to local anesthetics.
7. Patients with a history of treatment for chronic pain.
8. Previous history of breast surgery or other chest surgery.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours
  Visual Analog scale ≥6 using opioid (3mg morphine) VAS score is from 0 to 10 as 0 is no pain and 10 the wariest pain can ever experience
Visual Analog scale score postoperative | 24 hours
  Visual Analog scale≥4 using non-steroidal anti-inflammatory analgesic (ketorolac 30 mg) and VAS≥6 using opioid (3mg morphine) (0 mean no pain - 10 mean worset pain ever)

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | intraoperative
  total fentanyl consumption
Heart rate intraoperative | intraoperative
  ≥ 20 % of base line
Timing of first rescue analgesia | 24 hours
  first time patient needs analgesia

CONTACTS AND LOCATIONS:
Overall Officials: ahmed soliman, Principal Investigator — National Cancer Institute Cairo university
Locations (1):
- National cancer Insititute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No